CLINICAL TRIAL: NCT05538832
Title: Remote State Representation in Early Psychosis
Acronym: Rem-STEP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00020834; 5P50MH119569 (NIH)
Record Dates: First submitted 2022-08-05; First posted 2022-09-14 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Psychosis; Schizophrenia; Schizo Affective Disorder; Schizoaffective Disorder; Schizophreniform Disorders; Psychotic Disorders; Psychotic Mood Disorders; Psychoses, Affective; Psychosis Nos/Other; Schizophrenia Spectrum and Other Psychotic Disorders
Keywords: Cognitive Training; Remote; Online; Clinical Trial
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Affective Disorders, Psychotic; Schizophrenia Spectrum and Other Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The investigator will not know the treatment condition until the trial is completed. Participants will not be notified of which group they are assigned. The study coordinator will be aware of assignment but will not complete any outcomes assessments--these will be self-report.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Visual Perception Training (Experimental): Contains targeted visual perception exercises from BrainHQ's suite of cognitive exercises. This training paradigm is designed to improve state estimation processes at the perceptual input level.
  Interventions: Device: BrainHQ Computerized Cognitive Training - Visual Perception Training Paradigm
- Visual Cognitive Control Training (Experimental): Contains targeted visual cognitive control exercises from BrainHQ's suite of exercises. This training paradigm is designed to enhance state representation stability of visual information.
  Interventions: Device: BrainHQ Computerized Cognitive Training - Visual Cognitive Control Training Paradigm

INTERVENTIONS:
Device: BrainHQ Computerized Cognitive Training - Visual Perception Training Paradigm — The Cognitive Training is a program consisting of the follow set of exercises developed by Posit Science Corporation (BrainHQ) which is to be evaluated for Visual Perception Training: Visual Sweeps; Mind's Eye; Hawk Eye; and Divided Attention. Participants use a standard web browser on a broadband connected computer and go to the study web site. Participants perform multiple trials over the course of a session, with auditory/visual feedback and rewards to indicate if the trial was performed correctly or incorrectly. After each assigned session, the difficulty of the next session is updated to ensure that each participant is appropriately challenged.
  Arms: Visual Perception Training
Device: BrainHQ Computerized Cognitive Training - Visual Cognitive Control Training Paradigm — The Cognitive Training is a program consisting of the follow set of exercises developed by Posit Science Corporation (BrainHQ) which is to be evaluated for Visual Cognitive Control Training: Mind Bender; Divided Attention; Card Shark; and Freeze Frame. Participants use a standard web browser on a broadband connected computer and go to the study web site. Participants perform multiple trials over the course of a session, with auditory/visual feedback and rewards to indicate if the trial was performed correctly or incorrectly. After each assigned session, the difficulty of the next session is updated to ensure that each participant is appropriately challenged.
  Arms: Visual Cognitive Control Training

SUMMARY:
The purpose of this study is to examine state representation in individuals aged 18-30 who have been diagnosed with a psychotic illness, as well as young adults who do not have a psychiatric diagnosis. State Representation is our ability to process information about our surroundings. The investigators will complete some observational tests as well as a cognitive training clinical trial.

DETAILED DESCRIPTION:
The purpose of the current study is to investigate computationally-informed precision treatments to improve two forms of state representation dysfunction observed in psychosis: 1) Abnormal perceptual inputs that impair state estimation; or, 2) Reduced state representation stability that affects cognitive control, working memory, and behavioral outputs. We will test the effects of two forms of cognitive training: visual perception training or visual cognitive control training in individuals with early psychosis. Participants will have the option to complete all training and assessments entirely remotely. We will recruit both young adults who have been diagnosed with a psychosis spectrum illness (such as schizophrenia) as well as individuals without a history of psychosis to participate in this study.

Early psychosis can manifest low-level perceptual deficits (such as an abnormal mismatch negativity response); these perceptual abnormalities are observed in ~60% of individuals, where they are predictive of more severe disability at 12 month follow-up, consistent with multiple studies showing that perceptual input abnormalities, when present, have a widespread deleterious downstream impact. Psychotic disorders can also manifest deficits in working memory, consistent with dysfunctional state representation stability, seen in ~80% of patients. Thus, psychosis is heterogeneous in its underlying information processing pathology and clinical course, indicating a critical unmet need for precision treatment approaches.

We will address this unmet need by investigating the behavioral and neurophysiologic effects of a brief course of either visual perception training (designed to improve state estimation processes at the perceptual input level) or visual cognitive control training (designed to enhance state representation stability of visual information), in individuals with psychotic disorders such as schizophrenia, schizoaffective disorder, and bipolar disorder with psychosis. Because study visits may be conducted remotely, participants will be drawn from a national sample. Our goal is not to perform a treatment efficacy study comparing these two interventions. Rather, we seek to use predictions derived from basic and computational neuroscience to test the effects of neuroplasticity-based precision treatments targeting two distinct contributing information processing pathologies in psychosis, with the goal of improving state representation processes and cognition.

ELIGIBILITY:
INCLUSION CRITERIA

All Participants:

* Between the ages of 18-30 at the time of screening
* Fluent in spoken and written English, in that the participant learned to speak English before the age of 12 or is able to demonstrate fluency in conversation with study staff
* Has an outpatient status and no hospitalization for psychiatric reasons for at least 1 month prior to participant
* Has access to a computer with internet connection
* Has a United States address as permanent residence
* Estimated IQ at or above 70, as estimated by the cognitive assessments

Early Psychosis Participants:

* Diagnosis of one of the following conditions (confirmed via interview): schizophrenia; schizoaffective disorder; schizophreniform disorder; Psychosis not otherwise specified (NOS); major depressive disorder with psychotic features; bipolar disorder with psychotic features
* Willing to share contact with a clinical provider

EXCLUSION CRITERIA

All participants:

* History of severe substance use in the past 3 months (determined by interview)
* Unable to demonstrate capacity to consent to research, in the judgment of the study team
* Diagnosed with a neurological disorder that would impede participation in the study or would put the participant at additional risk by participating, in the opinion of the PI/CO-Is
* Previous clinically significant head injury or prolonged unconsciousness
* Significant cognitive training experience in the past 6 months
* Meets criteria for clinical risk of suicidal behavior.

Non-Psychosis participants:

* Meets DSM-5 criteria for a psychotic, bipolar, or autism spectrum disorder
* Has a family history (1st degree relative) of psychosis, bipolar, or autism spectrum disorders

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2022-07-27 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Performance of Dot Pattern Expectancy (DPX) Task Variant | Baseline, Immediately after the intervention, 5 month follow up
  The DPX task variant consists of a series of pattern sequences. One pattern is designated the "A" cue, and another the "X" cue, which requires one response (AX, 60-70% of trials, e.g. respond with the left button), while other sequences require a different response (AY or BX, 12-15% of trials each, or BY, 6-10% of trials, e.g. respond with the right button). Given the strong expectation that X's evokes a valid response, BX trials place demands on the fidelity (stability, memory) of the "B" cue state representation to overcome this tendency.
Change in Performance of Bandit Task Variant | Baseline, Immediately after the intervention, 5 month follow up
  This is a task variant that uses choice options (neutral images) that are rewarded probabilistically. The rewarded stimulus with the highest reward is changed over time. State learning associated with staying or switching stimuli too quickly (lose-switching) can be evaluated.

SECONDARY OUTCOMES:
Change in Test My Brain Neurocognitive Assessment performance: Global Cognition Z Score. | Baseline, Immediately after the intervention, 5 month follow up
  The investigators will examine global cognition scores from the Test My Brain neurocognitive battery. Z scores range from -5 to 5, with higher score indicating increased cognitive functioning.
Change in Test My Brain Neurocognitive Assessment performance: Verbal Pair Associates Memory Z Score | Baseline, Immediately after the intervention, 5 month follow up
  This subdomain of the TMB battery assesses verbal learning. Z scores range from -5 to 5, with higher score indicating increased functioning.
Change in Test My Brain Neurocognitive Assessment performance: Matrix Reasoning Z Score | Baseline, Immediately after the intervention, 5 month follow up
  This subdomain of the TMB battery assesses reasoning skills and also provides an IQ estimate. Z scores range from -5 to 5, with higher score indicating increased functioning.
Change in Test My Brain Neurocognitive Assessment performance: Multiracial Emotion Identification Z Score | Baseline, Immediately after the intervention, 5 month follow up
  This subdomain of the TMB battery is a social cognition test that assesses the ability to recognize emotions (happiness, sadness, anger, and fear). Z scores range from -5 to 5, with higher score indicating increased functioning.
Change in symptoms and functioning as indicated by Minnesota Symptom Severity Scale | Baseline, Immediately after the intervention, 5 month follow up
  This 29-item measure assesses symptoms in several domains such as anxiety, depression, sleep problems, somatic symptoms, and substance use. Scores range from 0 to 116, with a higher score indicating greater symptom severity.
Change in symptoms and functioning as indicated by the SANS/SAPS | Baseline, Immediately after the intervention, 5 month follow up
  The Scale for Assessment of Negative Symptoms (SANS, 25 items) and Scale for Assessment of Positive Symptoms (SAPS, 34 items) assess negative and positive symptoms of schizophrenia in a standardized interview. Scores on the SANS ranges from 0-125, and the SANS ranges from 0-170, with higher scores indicating increased symptom severity.
Change in symptoms and functioning as indicated by the BPRS | Baseline, Immediately after the intervention, 5 month follow up
  The Brief Psychiatric Rating Scale is a 24-item interview which assesses psychiatric symptoms. Scores on the BPRS rang from 24-168, with a higher score indicating increased symptom severity.
Change in symptoms and functioning as indicated by the GFS/GFR | Baseline, Immediately after the intervention, 5 month follow up
  The Global Functioning Social/Global Functioning Role scales provide a rating on a scale from 1-10 for social functioning and for role functioning, with higher scores indicating increased functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Demro, PhD, Principal Investigator — University of Minnesota Department of Psychiatry and Behavioral Sciences
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No